CLINICAL TRIAL: NCT02363582
Title: The Impact of a Prebiotics and Lactoferrin Containing Infant Formula on Stool Characteristics in Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang WU, MD, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SCMCIRB-K2013005
Record Dates: First submitted 2015-01-31; First posted 2015-02-16 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Infant Formula Intolerance
MeSH Terms: interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast fed (No Intervention): healthy term infants on exclusively breast feeding , enrollment age: 30-50days old
- Formula fed (Experimental): healthy term infants on exclusively formula fed , enrollment age: 30-50days old
  Interventions: Other: formula

INTERVENTIONS:
Other: formula — An infant formula contains prebiotics and lactoferrin
  Arms: Formula fed

SUMMARY:
Human milk (HM) is considered the gold standard nutrient for infants, which contains a lot of beneficial nutrients such as prebiotics and lactoferrin. Previous studies have shown that both prebiotics and lactoferrin play important roles in generating a bifidobacteria-dominated colonic microflora.The purpose of this study is to investigate the stool characteristics,acceptability, and gastrointestinal tolerance in term infants fed a starting infant formula supplemented with prebiotics and lactoferrin.

DETAILED DESCRIPTION:
Human milk (HM) is considered the gold standard nutrient for infants, which contains a lot of beneficial nutrients such as prebiotics and lactoferrin. Previous studies have shown that both prebiotics and lactoferrin play important roles in generating a bifidobacteria-dominated colonic microflora as well as the intestinal immune systems. The purpose of this study is to investigate the stool characteristics（including intestinal microbiota） acceptability, and gastrointestinal tolerance in infants fed a starting infant formula supplemented with prebiotics and lactoferrin, and compared these data with infants on exclusively breast feeding.

ELIGIBILITY:
Inclusion Criteria:

* full-term with a birth weight ≥2,500 g
* be in good health
* without symptoms of diarrhea, and had not received antibiotics for at least 1 week before enrollment
* exclusively fed by breast milk or infant formula

Exclusion Criteria:

* preterm infant
* with known diseases or currently taking medication drugs
* mixed feeding
* with symptoms of diarrhea
* received antibiotics within 1 week

Ages: 5 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
growth | 6 weeks
  Head circumferences and weight gain

SECONDARY OUTCOMES:
Gastrointestinal tolerance and safety | 6 weeks
  daily records of vomiting and stool characteristics; records of infection episodes and other adverse effects
intestinal microbiota | 6 weeks
  test the bacteria composition in baby stools by DNA sequencing technology

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, MD, Principal Investigator — Xin Hua Hospital
Locations (1):
- Xin Hua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No